CLINICAL TRIAL: NCT05541965
Title: The Effect of Reflexology and Pelvic Floor Muscle Exercises (Kegel) on Urinary Incontinence in MS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Afitap Ozdelikara, Associate Proffesor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Reflexology55
Record Dates: First submitted 2022-09-09; First posted 2022-09-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Reflexology; Urinary Incontinence
Keywords: Multiple sclerosis; Nurses; Complementary Therapies; Urinary Incontinence; Reflexology
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Median score distributions of the reflexology groups, ICIQ-SF, IQOL and ISI (Experimental)
  Interventions: Other: Reflexology and kegel exercises
- Median score distributions of the kegel groups, ICIQ-SF, IQOL and ISI (Active Comparator)
  Interventions: Other: Reflexology and kegel exercises
- Median score distributions of the control groups, ICIQ-SF, IQOL and ISI (Active Comparator)
  Interventions: Other: Reflexology and kegel exercises

INTERVENTIONS:
Other: Reflexology and kegel exercises — Reflexology is specific to a foot massage, and ıt can use different symptoms for patients.
  Kegel exercise is specific an activities and ıt can used for urinary incontinence

SUMMARY:
The research was carried out as experiment, control group, pretest-posttest model and single-blind. The population of the study consisted of MS patients who applied to OMU (Ondokuz Mayıs University) Neurology Service and Neurology Outpatient Clinic between March 2020 and February 2022. Fifteen patients who met the inclusion criteria were included in the study. Patients were divided into reflexology, pelvic floor muscle exercise and control groups. The control group was not intervened, only data collection tools were applied.

DETAILED DESCRIPTION:
The research was carried out as experiment, control group, pretest-posttest model and single-blind. The population of the study consisted of MS patients who applied to OMU (Ondokuz Mayıs University) Neurology Service and Neurology Outpatient Clinic between March 2020 and February 2022. Fifteen patients who met the inclusion criteria were included in the study. Patients were divided into reflexology, pelvic floor muscle exercise and control groups. The control group was not intervened, only data collection tools were applied.

reflexology intervention The reflexology application was carried out in a separate and quiet room, on a stretcher/bed where the patient could lie down, by adjusting the temperature so that they would not feel cold/sweaty. First, the feet were cleaned with a warm, damp cotton towel. Odorless, room temperature baby oil was used to provide lubricity during the reflexology application. The reflexology protocol was started with the right foot. First of all, rotation, vibration, etc. are applied to the ankle and ankle areas. relaxation techniques were applied for 2 minutes. Afterwards, reflexology massage was applied to the spinal cord, brain, pituitary areas, kidney, ureter and bladder areas with appropriate techniques. The session was concluded with solar plexus compression and relaxation maneuvers. The same protocol was applied in the left foot. Immediately after each reflexology session, the patient was allowed to drink 1 glass (200 ml) of water to accelerate the excretion of toxic products. Reflexology session was completed in 40 minutes for both feet. Foot reflexology was applied to the reflexology group twice a week (40 minutes for both feet) for a total of 4 weeks.

Pelvic floor muscle exercise (Kegel) application In the Kegel exercise group, the patients were taught the Kegel exercise at the first interview, and it was provided to be done under the guidance of the researcher. Afterward, they were asked to apply at least three times a day for four weeks, and a reminder SMS was sent to the patients daily.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS at least 6 months ago,
* Having an EDSS of <5,

Exclusion Criteria:

* To have wound on foots, varicose veins, etc. history of fractures causing loss of function, nail fungus,
* pregnancy,
* presence of acute infection
* To using any diuretic or incontinence medication,
* To have a curettage or pregnancy history in the last 6 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Index of severity incontinence (ISI) | 4 weeks
  The total score is between 0-12. A score of "0" indicates that there is no incontinence. The scale score is then categorized into 4 different levels of incontinence severity: 1-2: mild, 3-6: moderate, 8-9: severe, 10-12: very serious.
nternational Consultation on Incontinence Questionnaire Short Form(ICIQ-SF) | 4 weeks
  The scores that can be obtained from the scale range from 0 to 21; A low score indicates that urinary incontinence has little effect on quality of life, while a high score indicates that it affects the quality of life very much.
Incontinence quality of life (IQOL) | 4 weeks
  The total score ranges from 0 to 100. High scores indicate better quality of life than low scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Afitap ÖZDELİKARA, Samsun, Turkey (Türkiye)